CLINICAL TRIAL: NCT02849015
Title: Combination of Cryosurgery and NK Immunotherapy for Tumors in Transplanted Liver
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Shenzhen Hank Bioengineering Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK-liverTx
Record Dates: First submitted 2016-07-21; First posted 2016-07-29 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2018-07

CONDITIONS: Liver Tumor; Evidence of Liver Transplantation
Keywords: liver tumor; cryosurgery; NK immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cryosurgery

ARMS (2):
- Cryosurgery and NK immunotherapy (Experimental): In this group, the patients will receive liver cryosurgery first to destroy big tumors, then receive multiple NK immunotherapy (intensive treatment: 6 times in first 3 months; then interval treatment: once every 3 months). The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Device: Cryosurgery; Biological: NK immunotherapy
- Cryosurgery (Active Comparator): In this group, the patients will receive liver cryosurgery to destroy big tumors. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Device: Cryosurgery

INTERVENTIONS:
Device: Cryosurgery — Argon-helium cryosurgical system (percutaneous ablation under CT or ultrasound guidance)
Biological: NK immunotherapy — Natural killer cell(each treatment: about 10 billion cells transfusion in 3 times, i.v.)
  Arms: Cryosurgery and NK immunotherapy

SUMMARY:
The aim of this study is the safety and efficacy of cryosurgery plus natural killer(NK) immunotherapy to tumors in transplanted liver.

DETAILED DESCRIPTION:
By enrolling patients with tumors in transplanted liver adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of the combined therapy using cryosurgery and NK cells.

The safety will be evaluated by statistics of adverse reactions. The efficacy will be evaluated according to local relief degree, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* All standard therapies have failed according to NCCN guidelines or the patient refuses standard therapies after cancer recurrence
* Body tumor 1-6, the maximum tumor length < 5 cm
* KPS ≥ 70, lifespan > 6 months
* Platelet count ≥ 80×109/L，white blood cell count ≥ 3×109/L, neutrophil count ≥ 2×109/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 months

SECONDARY OUTCOMES:
Progress free survival（PFS） | 1 year
Overall survival（OS） | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jibing Chen, MD, PhD, Principal Investigator — Fuda Cancer Hospital, Guangzhou
Locations (1):
- Cancer Institute of Fuda cancer hospital, Guangzhou, Guangdong, China